CLINICAL TRIAL: NCT02417142
Title: Exenatide Weekly Injections as an Adjunctive Treatment in Patients With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Xiaoduo Fan, Xiaoduo Fan, MD, MPH, MS, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13T-005
Record Dates: First submitted 2015-04-10; First posted 2015-04-15 (Estimated); Results first posted 2021-06-15 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental (Experimental): Exenatide 2mg subcutaneous injection, once weekly
  Interventions: Drug: Exenatide
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Exenatide — Exenatide SQ 2mg/week for 24 weeks.
  Other Names: Bydureon
  Arms: Experimental
Drug: Placebo — Placebo SQ 1x/week for 24 weeks.
  Other Names: Control
  Arms: Placebo

SUMMARY:
This is a 24-week, randomized, double-blind, placebo-controlled trial of exenatide weekly injection (2mg per dose) as an adjunctive therapy in 70 schizophrenia subjects to examine exenatide's effects on negative symptoms and cognition.

DETAILED DESCRIPTION:
The specific aims include:

Primary aim:

1. Examine the efficacy of exenatide weekly injection in improving negative symptoms as measured by the Scale for the Assessment of Negative Symptoms (SANS) total score.

Secondary aims:

1. Examine the efficacy of exenatide in improving cognition as measured by the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) composite score.

Tertiary/Exploratory aims:

1. Examine exenatide's effect on schizophrenia symptoms as measured by the Positive and Negative Syndrome Scale (PANSS) total score.
2. Examine the efficacy of exenatide in improving social function as measured by the Instrumental Activities of Daily Living Scale (IADL) and the Heinrich Carpenter Quality of Life Scale (QLS).
3. Examine exenatide's effect on neuro-protection as measured by the change in hippocampal volume.
4. Examine exenatide's effects on inflammatory markers including serum levels of high sensitivity C-reactive Protein (CRP), Interleukin 6 (IL-6), and tumor necrosis factor (TNF-α).
5. Examine the potential moderator role of baseline serum levels of C-reactive Protein (CRP), Interleukin 6 (IL-6), tumor necrosis factor (TNF-α), and baseline hippocampal volume for exenatide's effects on negative and cognitive symptoms.
6. Examine the potential mediator role of changes from baseline in serum levels of C-reactive Protein (CRP), Interleukin 6 (IL-6), tumor necrosis factor (TNF-α), and hippocampal volume for exenatide's effects on negative and cognitive symptoms.
7. Examine the efficacy of exenatide in reducing body weight and improving glucose metabolism as measured by fasting plasma glucose and HbA1c.
8. Examine the safety and tolerability of exenatide as measured by changes in the side effects questionnaire (SEQ, SEQabbrev), EKG and vital signs

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 years
* diagnosis of schizophrenia or schizoaffective disorder
* stable dose of the current antipsychotic drug for at least one month
* well established compliance with outpatient treatment per treating clinician's judgment
* able to complete the cognitive assessment battery (must be English speaking)
* Female subjects will be eligible to participate in the study if they are of non-childbearing potential or of child-bearing potential and willing to practice appropriate birth control methods during the study

Exclusion Criteria:

* inability to provide informed consent
* current substance abuse
* psychiatrically unstable per treating clinician's judgment
* significant medical illnesses including uncontrolled hypertension, diabetes, seizure disorder, severe cardiovascular, cerebrovascular, pulmonary, or thyroid diseases
* currently on anti-inflammatory or immunosuppressant medication including oral steroids
* currently on sulfonylurea drugs (e.g. glyburide)
* history of chronic infection (including tuberculosis, HIV and hepatitis), malignancy, organ transplantation, blood dyscrasia, central nervous system demyelinating disorder, and any other known autoimmune or inflammatory condition
* pregnant or breastfeeding
* prisoners

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2020-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoduo Fan, MD, MPH, MS, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- UMass Medical School, Worcester, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Single-site study conducted at University of Massachusetts (UMass) Medical School. Subjects were recruited from UMass Memorial Healthcare facilities and ambulatory clinics in Worcester, MA.
Pre-assignment Details: Subjects who met DSM-IV (Diagnostic and Statistical Manual of Mental Disorders, 4th Edition) criteria for schizophrenia or schizoaffective disorder were enrolled in the study (see inclusion/exclusion criteria). Eligible subjects were randomly assigned to either the experimental or placebo group.
Groups:
- Experimental: (existing treatment) + (Drug)
  Intervention:
  Drug: Exenatide
  Exenatide: Exenatide 2mg/week subcutaneous injection for 24 weeks.
- Placebo: (existing treatment) + (Placebo)
  Intervention:
  Drug: Placebo
  Placebo: Placebo IM for 24 weeks.
Period: Overall Study
Arm/Group | Experimental | Placebo
Started | 35 | 35
Completed | 19 | 22
Not Completed | 16 | 13

BASELINE CHARACTERISTICS:
Groups:
- Experimental: (existing treatment) + (Drug)
  Intervention:
  Drug: Exenatide
  Exenatide: Exenatide IM 2mg/week for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Experimental | Placebo | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (12.3) | 43.9 (11.9) | 42.7 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 26 | 29 | 55
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 26 | 26 | 52
  Black/African American | 4 | 6 | 10
  Asian | 2 | 0 | 2
  Mixed | 1 | 3 | 4
  Unknown/Not reported | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35 | 35 | 70
Education [Mean (Standard Deviation); unit: years] | 12.9 (2.4) | 12.7 (2.1) | 12.8 (2.3)
Age of illness onset [Mean (Standard Deviation); unit: years] | 23.7 (8.3) | 24.6 (9.3) | 24.2 (8.8)
Duration of illness [Mean (Standard Deviation); unit: years] | 18.1 (12.2) | 18.9 (10.1) | 18.5 (11.2)
Schizophrenia [Count of Participants; unit: Participants] | 19 | 18 | 37
Schizoaffective disorder [Count of Participants; unit: Participants] | 16 | 17 | 33
Typical antipsychotic medication [Count of Participants; unit: Participants]
  Yes | 9 | 13 | 22
  No | 26 | 22 | 48
Atypical antipsychotic medication [Count of Participants; unit: Participants]
  Yes | 27 | 30 | 57
  No | 8 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Negative Symptoms as Measured by the Scale for the Assessment of Negative Symptoms (SANS) Total Score
Description: SANS measures negative symptoms on a 25-item, six point scale each (0-5; none-severe). Items are listed under five domains including affective flattening or blunting, alogia, avolition/apathy, anhedonia/asociality, and attention. The total possible score ranges from 0 to 125.
Time Frame: Baseline, Week 6, Week 12, Week 18 and Week 24
Population: 12 subjects in experimental arm withdrew or were lost to follow-up by week 24. 4 subjects in the experimental arm were removed from study by investigator by week 24.
  11 subjects in placebo arm withdrew or were lost to follow-up by week 24. 2 subjects in the placebo arm were removed from study by investigator by week 24.
  Reasons for removal include inpatient hospitalization, increase in depressive symptoms, elevated HbA1c, starting insulin therapy and repeatedly missing visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 35 | 35
score on a scale
  Baseline | 33.1 (12.9) | 34.1 (15.0)
  Week 6: number analyzed (Participants) | 30 | 25
  Week 6 | 34.1 (2.3) | 32.8 (11.8)
  Week 12: number analyzed (Participants) | 23 | 25
  Week 12 | 35.8 (13.0) | 34.5 (11.5)
  Week 18: number analyzed (Participants) | 22 | 23
  Week 18 | 36.1 (11.9) | 35.2 (10.2)
  Week 24: number analyzed (Participants) | 19 | 22
  Week 24 | 35.2 (13.3) | 35.0 (11.1)

2. Secondary Outcome: Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) Composite T-score
Description: The MATRICS Consensus Cognitive Battery (MCCB) measures cognition relevant to schizophrenia and related disorders. The MCCB consists of ten individually administered tests that measure cognitive performance in seven domains including speed of processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition. The raw scores from the ten tests are entered in the MCCB Computer Scoring Program software, which provides an age and gender-corrected T-score and percentile on the seven cognitive domains. A T-score of 50 +/- 10 represents a normative mean performance in each test. Accordingly, the criterion for assignment to cognitively normal-range group require an overall composite T-score from 40 to 60. These data points from baseline visit to week 24 will measure changes in cognition in addition overall cognitive ability compared to healthy individuals.
Time Frame: Baseline, Week 6, Week 12, Week 18, and Week 24.
Population: 12 subjects in experimental arm withdrew or were lost to follow-up by week 24. 4 subjects in the experimental arm were removed from study by investigator by week 24.
  11 subjects in placebo arm withdrew or were lost to follow-up by week 24. 2 subjects in the placebo arm were removed from study by investigator by week 24.
  Reasons for removal include inpatient hospitalization, increase in depressive symptoms, elevated HbA1c, starting insulin and repeatedly missing visits during study period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 35 | 35
score on a scale
  Baseline | 26.9 (17.2) | 24.7 (12.6)
  Week 6: number analyzed (Participants) | 30 | 25
  Week 6 | 27.3 (17.3) | 27.2 (15.4)
  Week 12: number analyzed (Participants) | 23 | 25
  Week 12 | 28.4 (17.3) | 28.1 (16.2)
  Week 18: number analyzed (Participants) | 22 | 23
  Week 18 | 28.7 (18.1) | 32.2 (15.1)
  Week 24: number analyzed (Participants) | 19 | 22
  Week 24 | 31.2 (16.5) | 33.9 (14.4)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Experimental | Placebo
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 29/35 | 27/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental (N=35) | Placebo (N=35)
Bump at injection site (Skin and subcutaneous tissue disorders) | 17 | 0
Headache (General disorders) | 9 | 10
Heartburn (Gastrointestinal disorders) | 5 | 8
Constipation (Gastrointestinal disorders) | 5 | 8
Itchiness at injection site (Skin and subcutaneous tissue disorders) | 8 | 0
Nausea (General disorders) | 4 | 2
Irritability/anxiety (Psychiatric disorders) | 7 | 3
Vomiting (Gastrointestinal disorders) | 2 | 6
Diarrhea (Gastrointestinal disorders) | 3 | 3
Dizziness (General disorders) | 3 | 3
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Fatigue (General disorders) | 3 | 2
Indigestion (Gastrointestinal disorders) | 3 | 1
Chest pain (Cardiac disorders) | 3 | 0
Hunger (General disorders) | 2 | 2
Suicidal Ideation (Psychiatric disorders) | 2 | 3
Decreased appetite (General disorders) | 2 | 1
Sedation (General disorders) | 2 | 1
Blurry vision (Eye disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-11-30): https://cdn.clinicaltrials.gov/large-docs/42/NCT02417142/Prot_002.pdf
  • Statistical Analysis Plan (2019-11-30): https://cdn.clinicaltrials.gov/large-docs/42/NCT02417142/SAP_001.pdf